CLINICAL TRIAL: NCT00124488
Title: Comparison of Tomotherapy Versus Intensity-modulated Step-and-shoot and Conventional Radiation Treatment Plans for Patients With Locally-advanced Squamous Cell Carcinoma of the Cervix
Status: Completed | Type: Observational
Sponsor: Alberta Health services (Other)
Organization: AHS Cancer Control Alberta (Other)
Other Study IDs: NA-15-0004
Record Dates: First submitted 2005-07-26; First posted 2005-07-28 (Estimated); Last update posted 2011-12-09 (Estimated); Status verified 2011-12

CONDITIONS: Cervix Neoplasm
Keywords: radiotherapy planning; computer assisted radiotherapy; conformal
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective

INTERVENTIONS:
Device: Tomotherapy Treatment Planning

SUMMARY:
Standard treatment for non-operable cervix cancer is radiation and chemotherapy. This treatment combination can result in significant radiation side-effects involving the bladder, small bowel and rectum. To improve results with radiation/chemotherapy, higher radiation doses have been tried for cervix cancer patients. Results from using higher radiation doses show that cervix tumours may be better controlled, but the radiation side-effects are worsened. Intensity modulated radiotherapy (IMRT) and Tomotherapy are new radiation planning and delivery technologies which may allow for delivery of higher radiation doses with less damage to normal organs. The purpose of this project is to determine whether or not IMRT and/or Tomotherapy technology can produce radiation plans that deliver higher doses of radiation to the tumor and lower doses to normal organs when compared to standard radiation plans. The results from this project will provide the basis for possibly treating future cervix cancer patients with Tomotherapy and providing them with improved cure rates along with decreased rates of radiation side effects. No patients will be treated on this protocol, as the investigators plan to only compare radiation dose calculations from different treatment plans created for test cervix cancer cases. There will be absolutely no patient contact in this protocol.

DETAILED DESCRIPTION:
Background Information:

The addition of concurrent chemotherapy to radiotherapy (RT) for locally-advanced cervix cancer has improved patient outcomes, but treatments are associated with significant rates of radiotherapy (RT)-related toxicities. Plus, the disease-free and overall survival benefits conferred by concurrent chemotherapy appear to be most prominent in patients with earlier stage disease. Limits to RT for cervix cancer which can impact patient outcomes are overall treatment time and RT dose. Attempts to overcome these limits have been made in trials using altered RT fractionation schemes. Promising rates of local control reported in these trials are offset by excessive rates of acute and late RT-related toxicities.

Intensity-modulated radiotherapy (IMRT) is innovative RT planning and delivery technology with the ability to vary the intensity of radiation across a beam, allowing for increased conformity of RT dose around target volumes along with decreased dose delivered to normal structures. Tomotherapy uses an intensity-modulated beam which rotates around the patient as the patient is being translated longitudinally through the gantry and features the ability to acquire megavoltage CT (MVCT) images of target structures at each treatment. It is thought that Tomotherapy can plan and deliver more conformal RT with the added advantage of daily assessment of target and critical structure position via MVCT imaging.

Experience with using IMRT for cervix cancer is sparse. Reports of treating pelvic nodal targets in small numbers of selected cervix cancer patients with IMRT suggests that the treatments are tolerable and associated with decreased incidences of acute and late RT-related toxicities compared with a similar patient cohort treated with conventional RT technologies. Currently, there is no published report of using Tomotherapy to plan or deliver RT using conventional or altered fractionation for cervix cancer patients.

The limitations of overall treatment time and the maximal dose of RT that can be safely delivered to the pelvis targets make cervical carcinoma a tumor in which Tomotherapy can potentially improve the therapeutic ratio. Tomotherapy's ability to deliver more conformal RT to target structures and minimize dose to normal structures may allow for delivery of altered fractionation radiation plans for cervix cancer with acceptable rates of RT-related toxicities. Tomotherapy allows for delivery of differential daily doses of RT to target volumes that lie within larger target volumes which in effect delivers a simultaneous integrated boost (SIB) to areas of gross disease which lie within a larger volume at risk for harbouring micrometastases. Delivery of the boost dose of radiation in a simultaneous as opposed to sequential fashion decreases the overall RT treatment time which theoretically reduces the effects of accelerated tumor cell repopulation. Delivering higher doses per fraction to areas of gross disease would theoretically increase the radiobiologic enhancement effects of concurrent cisplatin chemotherapy.

Tomotherapy represents a key advance in radiotherapy planning and delivery technology. Its potential dosimetric and radiobiologic advantages over standard radiotherapy technologies need evaluation in properly-conducted clinical trials. Prior to the initiation of such trials, it must be shown that Tomotherapy plans at least have dosimetric advantages over conventional plans.

Objective:

To compare radiotherapy (RT) plans created for locally-advanced cervix cancer cases using Tomotherapy, conventional computed tomography-based methods and step-and-shoot intensity-modulated methods.

Study Design:

Pre-treatment planning computed tomography scans of ten previously-treated cervix cancer patients will be used. All identifying patient data on these CT image sets will be completely removed. Three RT plans will be created for case: Tomotherapy, step-and-shoot IMRT, and conventional. The University Medical Centre in Utrecht, The Netherlands has implemented IMRT into clinical management of cervical cancer and the Gynecologic Oncology group there has graciously agreed to collaborate on this project by creating optimized step-and-shoot IMRT plans on our ten test cases. The anonymous CT image sets will be stored on data discs which will be sent via bonded courier to the University Medical Centre in Utrecht, The Netherlands for generation of step and shoot IMRT plans. Data to be calculated and collected from all plans include: dose-volume histograms (DVH's) for all target volumes and critical structures. Tumor Control Probability for targets and Normal Tissue Complication Probability for critical structures will be calculated. RT plans created on this protocol will only be used for dose and biophysical model calculation comparisons; no plan will be used to deliver actual radiation treatments to any patient. There will be absolutely no patient contact or interaction on this protocol.

Future Directions:

The investigators anticipate that results from this study will confirm the hypothesis that Tomotherapy plans incorporating a simultaneous integrated boost for cervix cancer will provide superior target volume coverage and normal critical structure avoidance when compared with step-and-shoot IMRT and conventional plans. Such confirmation will provide the basis to proceed with efforts to improve target and normal structure delineation for Tomotherapy treatment planning of cervix cancer using MRI-based planning. Ultimately, we plan to initiate phase I/II trials using MRI-based Tomotherapy planning and delivery techniques for cervix cancer patients. Incorporation of RT dose escalation and monitoring of treatment response with biologic imaging techniques for cervix cancer patients treated with Tomotherapy are other future potential areas of investigation.

ELIGIBILITY:
Inclusion Criteria:

* Squamous cell cervix cancer
* Undergone planning computed tomography (CT) scan for radiotherapy planning
* Treated with chemoradiotherapy

Exclusion Criteria:

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: primary care clinic
Sampling Method: Non-Probability Sample
Enrollment: 10
Dates: Start 2005-06; Study Completion 2005-11

CONTACTS AND LOCATIONS:
Overall Officials: Don Yee, MD, Principal Investigator — AHS Cancer Control Alberta
Locations (1):
- Cross Cancer Institute, Edmonton, Alberta, Canada

REFERENCES:
- [Background] Thomas GM. Concurrent chemotherapy and radiation for locally advanced cervical cancer: the new standard of care. Semin Radiat Oncol. 2000 Jan;10(1):44-50. doi: 10.1016/s1053-4296(00)80020-x. PMID 10671658
- [Background] Girinsky T, Rey A, Roche B, Haie C, Gerbaulet A, Randrianarivello H, Chassagne D. Overall treatment time in advanced cervical carcinomas: a critical parameter in treatment outcome. Int J Radiat Oncol Biol Phys. 1993 Dec 1;27(5):1051-6. doi: 10.1016/0360-3016(93)90522-w. PMID 8262826
- [Background] Fyles A, Keane TJ, Barton M, Simm J. The effect of treatment duration in the local control of cervix cancer. Radiother Oncol. 1992 Dec;25(4):273-9. doi: 10.1016/0167-8140(92)90247-r. PMID 1480773
- [Background] Petereit DG, Sarkaria JN, Chappell R, Fowler JF, Hartmann TJ, Kinsella TJ, Stitt JA, Thomadsen BR, Buchler DA. The adverse effect of treatment prolongation in cervical carcinoma. Int J Radiat Oncol Biol Phys. 1995 Jul 30;32(5):1301-7. doi: 10.1016/0360-3016(94)00635-X. PMID 7635769
- [Background] Perez CA, Grigsby PW, Chao KS, Mutch DG, Lockett MA. Tumor size, irradiation dose, and long-term outcome of carcinoma of uterine cervix. Int J Radiat Oncol Biol Phys. 1998 May 1;41(2):307-17. doi: 10.1016/s0360-3016(98)00067-4. PMID 9607346
- [Background] Kavanagh BD, Gieschen HL, Schmidt-Ullrich RK, Arthur D, Zwicker R, Kaufman N, Goplerud DR, Segreti EM, West RJ. A pilot study of concomitant boost accelerated superfractionated radiotherapy for stage III cancer of the uterine cervix. Int J Radiat Oncol Biol Phys. 1997 Jun 1;38(3):561-8. doi: 10.1016/s0360-3016(97)89484-9. PMID 9231680
- [Background] MacLeod C, Bernshaw D, Leung S, Narayan K, Firth I. Accelerated hyperfractionated radiotherapy for locally advanced cervix cancer. Int J Radiat Oncol Biol Phys. 1999 Jun 1;44(3):519-24. doi: 10.1016/s0360-3016(99)00043-7. PMID 10348280
- [Background] Viswanathan FR, Varghese C, Peedicayil A, Lakshmanan J, Narayan VP. Hyperfractionation in carcinoma of the cervix: tumor control and late bowel complications. Int J Radiat Oncol Biol Phys. 1999 Oct 1;45(3):653-6. doi: 10.1016/s0360-3016(99)00245-x. PMID 10524419
- [Background] Nutting C, Dearnaley DP, Webb S. Intensity modulated radiation therapy: a clinical review. Br J Radiol. 2000 May;73(869):459-69. doi: 10.1259/bjr.73.869.10884741.